CLINICAL TRIAL: NCT03961373
Title: Standard Versus Super-extended Lymphadenectomy After Neo-adjuvant Chemotherapy for Gastric Cancer
Acronym: Neo-D2plus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Franco Roviello, Full Professor, Clinical Research, University of Siena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neo-D2plus trial
Record Dates: First submitted 2019-03-12; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Locally Advanced Gastric Cancer
MeSH Terms: interventions — Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Group (Active Comparator): Neoadjuvant chemotherapy + surgical gastrectomy with D2 lymphadenectomy
  Interventions: Procedure: Gastrectomy with D2 lymphadenectomy
- Experimental Group (Experimental): Neoadjuvant chemotherapy + surgical gastrectomy with D2plus lymphadenectomy
  Interventions: Procedure: Gastrectomy with D2plus lymphadenectomy

INTERVENTIONS:
Procedure: Gastrectomy with D2 lymphadenectomy — Patients who are assigned to the neoadjuvant chemotherapy+ surgical D2 treatment group will undergo either subtotal or total gastrectomy, depending on the location of the primary tumour. Standardized D2-lymph node dissection is required with specific information about lymph node stations.
  Arms: Standard Group
Procedure: Gastrectomy with D2plus lymphadenectomy — Patients who are assigned to the neoadjuvant chemotherapy + surgical D2+ extended lymphadenectomy treatment group will undergo either subtotal or total gastrectomy, depending on the location of the primary tumour. Standardized D2+ lymph node dissection plus resection of stations 8p, 12p, 13, 14v, 16a2/b1 is required with specific information about lymph node stations.
  Arms: Experimental Group

SUMMARY:
In this study the patients with histological evidence of adenocarcinoma of the stomach will be screened and, if eligible, submitted to neo-adjuvant chemotherapy (NAC). After conclusions of NAC and obtaining informed consent, they will be registered and randomized to receive surgical D2 vs. D2plus lymphadenectomy.

DETAILED DESCRIPTION:
This is a prospective multi-centre phase III, two-group, randomized and controlled trial designed to prove superiority of the experimental treatment arm (neo-adjuvant chemotherapy and super-extended lymphadenectomy).

The trial population consists of patients who have histologically confirmed adenocarcinoma of the stomach with locally advanced primary tumour and no evidence of distant metastases (stage IIA-IIIC gastric cancer). The lymph node clinical metastases, before neo-adjuvant chemotherapy, must be limited to the first and second compartments (stations 1-12).

STANDARD GROUP: Neoadjuvant chemotherapy + surgical gastrectomy with D2 lymphadenectomy.

Patients who are assigned to neoadjuvant chemotherapy+ surgical D2 treatment group will undergo either subtotal or total gastrectomy, depending on the location of the primary tumour. Standardized D2-lymph node dissection is required with specific information about lymph node stations.

EXPERIMENTAL GROUP: Neoadjuvant chemotherapy + surgical gastrectomy with D2plus lymphadenectomy.

Patients who are assigned to neoadjuvant chemotherapy + surgical D2plus extended lymphadenectomy treatment group will undergo either subtotal or total gastrectomy, depending on the location of the primary tumour. Standardized D2 lymph node dissection plus resection of stations 8p, 12b/p, 13, 14v, 16a2/b1 is required with specific information about lymph node stations.

In both groups, surgical treatment should be performed within 4-6 weeks after the end of the last cycle of NAC.

The primary objective of this study is to compare overall and cancer-related survival between D2 and D2+ lymphadenectomy following neo-adjuvant chemotherapy for resectable gastric cancer.

In addition, response to chemotherapy, resection rate, quality of life, complications attributable to surgical intervention / side effects of chemotherapy and the duration of hospitalization will be evaluated.

Sample size estimation was performed, to detect the minimum number of patients to be recruited in each arm. A two-sided log rank test with an overall sample size of 539 subjects, of which 270 are in group 1 and 269 are in group 2.

Data will be analyzed using SPSS software. Level of significance will be defined as 5%.

The trial will be open for recruitment from October 2018 to September 2023.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 18 years
* IIA-IIIC histologically proven primary gastric adenocarcinoma, before the treatment with NAC. Not including gastro-oesophageal junction/cardia carcinoma but only Siewert 3, without any previous treatment (surgery and / or chemotherapy) for this diagnosis
* Lack in CT scan of following:

  1. Mediastinal lymph nodes
  2. Lung metastases
  3. Peritoneal metastases
  4. Liver metastases
  5. Pleural effusion, ascites
  6. Metastases to para-aortic lymph nodes No 16a2/b1
  7. Metastases to lymph nodes located in the "posterior" area (8p, 12 b/p, 13)
  8. Extra-regional lymph node metastases
* ECOG performance status ≤ 2
* No prior radio- or chemotherapy conflicting with the treatment of gastric cancer
* No oesophageal invasion, or invasion <=3cm
* Negative peritoneal washing cytology findings and no peritoneal metastases in staging laparoscopy
* No gastric stump cancer
* No signs of cervical and subclavear lymph nodes or distal metastases
* Patient's consent form obtained, signed and dated before beginning specific protocol procedures
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Exclusion Criteria:

* Contraindications for any sort of appropriate chemotherapy according to local standards
* Linitis plastica
* Second uncontrolled malignant tumour (synchronous or metachronous (last 5 years) other than Cis or mucosal cancer
* Neoplasms involving the esophago-gastric junction (Siewert types I and II)
* Expected unresectability after neo-adjuvant treatment or progression in metastases
* Emergency surgery due to bleeding or perforation
* Uncontrolled infections
* Other serious underlying medical conditions that could impair the ability of the patient to participate in the study
* Pregnant or lactating women
* Significant neurologic or psychiatric disorders
* Severe cardiac illness (NYHA class IV)
* Under treatment of systemic steroids
* Participation in any other clinical trial that might interfere with the results of this trial
* Lack of compliance
* Inability to fill in questionnaires (insufficient command of language, dementia, lack of time)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival analysis | This outcome measure will be estimated from the time of randomization to the date of death or last follow up visit, assessed approximately 5 years after the disease diagnosis.
  Overall survival analysis will be analysed during follow up visits

SECONDARY OUTCOMES:
Recurrence free-survival | This outcome measure will be estimated from the time of randomization to the date of recurrence, assessed approximately 5 years after the disease diagnosis.
  That part will also be analysed during follow up visits. The recurrence has to be documented in radiological, endoscopic or pathological examination, when possible.
Post-operative morbidity | This outcome measure will be assessed approximately 3 month after the operation date.
  Severity of post-operative complications will be analysed using Clavien-Dindo classification
Post-operative mortality | Within 30 days from operation or during the hospital stay
  Deaths after surgery
R0 resection | This outcome measure will be assessed approximately 3 month after the operation date.
  Absence of microscopic (R1) or macroscopic (R2) residual tumor after surgery
Percentage of completion of protocol treatment | This outcome measure will be assessed approximately 12 month after the date of enrollment.
  Percentage of patients who will complete the protocol treatment, including adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Franco Roviello, Principal Investigator — University of Siena
Locations (1):
- General and Surgical Oncology Department, University of Siena, Siena, Italy